CLINICAL TRIAL: NCT00217555
Title: Phase II Trial for the Treatment of Recurrent or Persistent Platinum-Refractory Ovarian, Fallopian Tube, or Primary Peritoneal Cancer With Gemcitabine and Topotecan
Brief Title: Gemcitabine and Topotecan in Treating Patients With Recurrent or Persistent Ovarian, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: PSOC 1901; PSOC-1901; GSK-PSOC-1901; PSOC-IRB-5320; LILLY-PSOC-1901; CDR0000441309 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Gemcitabine; Topotecan

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with topotecan works in treating patients with recurrent or persistent ovarian, fallopian tube, or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the nature and degree of toxicity of gemcitabine and topotecan in patients with recurrent or persistent platinum-refractory ovarian, fallopian tube, or primary peritoneal cavity cancer.
* Determine the response rate in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.

Secondary

* Determine the duration of progression-free survival and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes and topotecan IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses beyond documentation of CR.

Quality of life is assessed at baseline, on day 1 of courses 2, 4, and 6, and then at 1 year.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 36-45 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ovarian, fallopian tube, or primary peritoneal cavity cancer
* Recurrent or persistent platinum-refractory disease, as defined by 1 of the following:

  * Progressive disease while on a platinum compound
  * Persistent clinically measurable disease with best response as stable disease at the completion of ≥ 6 courses of therapy
  * Recurrent disease within 6 months after completion of therapy
* Measurable or evaluable disease

  * Evaluable disease, defined as CA 125 ≥ 100 U/mL (confirmed by 2 blood tests)
  * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI, OR ≥ 10 mm by spiral CT scan

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN
* Creatinine clearance > 50 mL/min

Other

* No clinically significant infection
* No other severe medical condition that would preclude study treatment
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix or breast

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* Prior gemcitabine or topotecan allowed provided disease is not refractory to either drug
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* At least 3 weeks since prior radiotherapy and recovered

Surgery

* Recovered from recent prior surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-07; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Toxicity
Response rate
Quality of life

SECONDARY OUTCOMES:
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Goff, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Medicine, Seattle, Washington, United States

REFERENCES:
- [Result] Goff BA, Holmberg LA, Veljovich D, Kurland BF; Puget Sound Oncology Consortium. Treatment of recurrent or persistent platinum-refractory ovarian, fallopian tube or primary peritoneal cancer with gemcitabine and topotecan: a phase II trial of the Puget Sound Oncology Consortium. Gynecol Oncol. 2008 Aug;110(2):146-51. doi: 10.1016/j.ygyno.2008.04.037. Epub 2008 Jun 6. PMID 18538834